CLINICAL TRIAL: NCT01434901
Title: The Effects of Bethanechol, a Muscarinic Agonist, on Plasma Insulin, Glucagon, and Glucose Levels in Humans With and Without Type 2 Diabetes Mellitus
Brief Title: The Effects of Bethanechol on Glucose Homeostasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 08-0861C; 1R01DK088126-01 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-09-15 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Blood Sugar; Xenin-25; GIP; Muscarinic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Bethanechol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal Glucose Tolerance (Experimental): Healthy individuals exhibiting plasma glucose levels less than 140mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Bethanechol (25 mg); Drug: Bethanechol (50 mg); Drug: Bethanechol (100 mg)
- Impaired Glucose Tolerance (Experimental): Healthy individuals exhibiting plasma glucose levels between 140 and 199 mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Bethanechol (25 mg); Drug: Bethanechol (50 mg); Drug: Bethanechol (100 mg)
- Type 2 Diabetes Mellitus (Experimental): Healthy individuals exhibiting plasma glucose levels greater than 150 mg/dL under fasting conditions OR greater than 199 mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Bethanechol (25 mg); Drug: Bethanechol (50 mg); Drug: Bethanechol (100 mg)

INTERVENTIONS:
Drug: Placebo — A placebo will be taken by mouth 1 hour before ingestion of a mixed meal.
Drug: Bethanechol (25 mg) — 25 mg of Bethanechol will be taken by mouth 1 hour before ingestion of a mixed meal
Drug: Bethanechol (50 mg) — 50 mg of Bethanechol will be taken by mouth 1 hour before ingestion of a mixed meal
Drug: Bethanechol (100 mg) — 100 mg of Bethanechol will be taken by mouth 1 hour before ingestion of a mixed meal

SUMMARY:
Xenin-25 and glucose-dependent insulinotropic polypeptide (GIP) are hormones produced in the intestine that are released into the blood immediately after ingestion of a meal. Together, these 2 hormones increase insulin release and reduce blood glucose levels. Xenin-25 works by increasing acetylcholine release in pancreatic islets. This study will determine if a Bethanechol, a drug that is similar to acetylcholine, also increases insulin release and reduces blood glucose levels after ingestion of a mixed meal.

DETAILED DESCRIPTION:
Each eligible participant will be administered an oral glucose tolerance test (OGTT) so he/she can be assigned to the group with normal glucose tolerance (NGT), impaired glucose tolerance (IGT) which is between normal and diabetic, or type 2 diabetes mellitus (T2DM). Each study subject will then be administered a meal tolerance test (MTT) on 4 separate occasions. For the MTT, a liquid meal (Boost Plus) will be ingested following an overnight fast. A placebo or Bethanechol (25 mg, 50 mg, or 100 mg) will taken by mouth 1 hour before ingestion of the meal. Blood samples will be collected before and during the MTT for the measurement of glucose, insulin, C-peptide, and glucagon levels.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65. No minors will be studied.
* Individuals must be able to consent for their own participation (no mental impairment affecting cognition or willingness to follow study instructions).
* Healthy volunteers with no clinical evidence of T2DM (see below).
* Otherwise healthy volunteers that have impaired glucose tolerance (see below).
* Otherwise healthy volunteers with Diet Controlled T2DM (see below).
* Otherwise healthy volunteers with T2DM that take oral agents only and if the subject's pre-existing oral anti-diabetic agents can be safely discontinued for 48 hours prior to Oral Glucose Tolerance Test.
* Otherwise healthy volunteers with T2DM who do not use insulin for blood glucose control.
* Persons with HbA1c ≤ 9%.
* Women of childbearing potential must be currently taking/using a method of birth control that is acceptable to the investigators. A pregnancy test will be done at the beginning of each visit. Any woman with a positive pregnancy test will be removed from the study.

Exclusion Criteria:

* <18years of age or >65 years of age
* Lacks cognitive ability to sign the consent &/or follow the study directions for themselves
* Women unwilling to comply with using an acceptable method of contraception during the course of the study, or who are currently breast-feeding.
* Any subject whose screening HbA1c is >9.0%
* Type 2 diabetes requiring the use of supplemental insulin @ home
* Volunteers with a history of Acute Pancreatitis
* Volunteer with a history of Chronic Pancreatitis and/or risk factors for chronic pancreatitis including hypertriglyceridemia (triglycerides >400mg/ml) hypercalcemia (blood calcium level >11.md/dl) and/or the presence of gallstones.
* Volunteers with a history of gastrointestinal disorders, particularly related to gastric motility/emptying such as gastric bypass, documented gastro-paresis in diabetic volunteers.
* Volunteers with a history of cancer. Exception: skin cancer.
* Diabetics that have the potential to have a low blood sugar without them being aware that their blood sugar is low (hypoglycemia unawareness).
* Known heart, kidney. liver or pancreatic disease requiring medications.
* Unwillingness to allow blood glucose level adjustment (if needed) with IV insulin.
* Subjects with hyperthyroidism, coronary artery disease, peptic ulcer, asthma, chronic bronchitis, or COPD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2014-07-07 (Actual); Study Completion 2014-07-07 (Actual)

PRIMARY OUTCOMES:
The effects of Bethanechol on insulin secretion rates | 3 years
  Insulin secretion rates (pmoles/min) will be calculated by deconvolution of plasma C-peptide levels. The investigators will then determine if post-prandial insulin secretion rates are greater following administration of Bethanechol compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Burton M Wice, PhD, Principal Investigator — Washington University School of Medicine; Dominic Reeds, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Chowdhury S, Wang S, Dunai J, Kilpatrick R, Oestricker LZ, Wallendorf MJ, Patterson BW, Reeds DN, Wice BM. Hormonal Responses to Cholinergic Input Are Different in Humans with and without Type 2 Diabetes Mellitus. PLoS One. 2016 Jun 15;11(6):e0156852. doi: 10.1371/journal.pone.0156852. eCollection 2016. PMID 27304975